CLINICAL TRIAL: NCT06579079
Title: A Hybrid Type III Implementation-effectiveness Trial to Improve Implementation and Participation of Universal School Meals (USM)
Brief Title: Improving Participation in Universal School Meals (USM)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: The School District of Philadelphia (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Gabriella McLoughlin, Assistant Professor, Temple University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: #28959
Record Dates: First submitted 2024-07-08; First posted 2024-08-30 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Food Deprivation; Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implementation Strategy - Intervention Condition (Experimental): Schools in the intervention condition will be assigned to receive coaching and logistical support to develop and tailor an implementation strategy across 1 academic year. This strategy will then be implemented gradually and in the following academic years (2- year pilot).
  Interventions: Other: Implementation Mapping
- Waitlist Control (Active Comparator): Schools in the waitlist control will wait 1 academic year before developing and testing an implementation strategy (1-year pilot)
  Interventions: Other: Waitlist Comparison - Implementation Mapping

INTERVENTIONS:
Other: Implementation Mapping — Implementation mapping is a stakeholder-driven process whereby researchers and practitioners work together to develop an implementation strategy.
  Arms: Implementation Strategy - Intervention Condition
Other: Waitlist Comparison - Implementation Mapping — Implementation mapping is a stakeholder-driven process whereby researchers and practitioners work together to develop an implementation strategy. Participating schools receiving this treatment will wait one year before developing an implementation strategy for testing.
  Arms: Waitlist Control

SUMMARY:
The purpose of this study is to assess the impact of an implementation strategy on participation in Universal School Meals (USM).

DETAILED DESCRIPTION:
The purpose of this cluster randomized trial is to test the effectiveness of an implementation strategy on implementation and student health outcomes of universal school meals (USM). This will be completed by developing and tailoring of an implementation strategy and testing its effectiveness though a cluster randomized design. Primary implementation outcomes of this trial are acceptability, cost, feasibility, penetration, and sustainability. Secondary student health outcomes are changes in diet quality (district-wide survey for students), food insecurity (USDA 6-item screener), and weight status. Exploratory descriptive models will be run to assess differences between intervention and control schools. To provide evidence for approaches in adolescents at highest risk for poor dietary intake, food security, and obesity risk, racial and ethnic minority adolescents from the School District of Philadelphia will comprise the majority of the sample. The principal investigator has just completed a year-long needs assessment with 8 schools across the district. We will aim to recruit 4 schools to be randomized to 1 of 2 conditions. Recruitment is underway, final recruitment details will be added once randomization is complete. From these schools, we aim to randomize (2 intervention; 2 waitlist comparison) for the development and tailoring of an implementation strategy. At baseline and throughout the 2-year trial period, we aim to collect interview data and surveys, and analyze data on diet quality, food security, and weight status.

ELIGIBILITY:
Inclusion Criteria:

* An elementary/middle or high school within the School District of Philadelphia (SDP) that provides free breakfast and lunch to students
* School is willing to be randomized to either a treatment or waitlist comparison condition
* School has a team of teachers, administration, and food service staff who are willing to complete interviews and surveys for data collection
* School has valid data for student Body Mass Index, meal participation, and food insecurity (parent reported).
* Students currently enrolled in a SDP elementary/middle/high school
* Students willing to participate in an interview and complete surveys
* Students have participated in school meals in the last year.

Exclusion Criteria:

* Charter schools and private schools
* Students not enrolled in school full time; students under 11 years of age.

Ages: 11 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
School Meal Participation | Throughout study completion
  Counts to calculate number of students who participate in breakfast and lunch each day will be generated and totaled for each school.
Qualitative Interviews | 1 year
  Focus group interviews with students, parents, teachers, administration, and food service staff.
Implementation Mapping Self-Assessment | 1 year
  Self-assessment to document fidelity to implementation mapping procedures.
Implementation Cost Measure | 1 Year
  A survey developed through stakeholder interviews to calculate costs of implementation will be completed by schools.
Implementation Outcomes Surveys | 1 Year
  Implementation outcomes of perceived acceptability, feasibility, and sustainability of the implementation strategy will be assessed through surveys completed by school stakeholders

SECONDARY OUTCOMES:
Height | Baseline and 1 year
  Student height (feet, inches) is collected by school nurses and other professionals in the school district. These data are a secondary outcome to implementation outcomes.
Food Insecurity | Baseline and 1 year
  The United States Department of Agriculture (USDA) 6-item food screening questionnaire is administered to parents across the district. These data are a secondary outcome to implementation outcomes.
Dietary Behaviors | Baseline and 1 year
  Students complete a survey each year which records their nutrition behaviors such as fruit and vegetable consumption, sugar-sweetened beverages, and other key behaviors. These data are a secondary outcome to implementation outcomes.
Student Weight | Baseline and 1 year
  Student weight (pounds) is collected by school nurses and other professionals in the school district. These data are a secondary outcome to implementation outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data elements: 1) Individual linked integrated database containing up to ~1000 records from the School District of Philadelphia from 2024-2027; 2) up to ~100 interview recordings and transcripts conducted with students in middle (6-8) and high (9-12) school grades, teachers, food service staff/personnel, administrators, and other staff; 3) up to ~30-50 survey entries to capture implementation outcomes of acceptability, feasibility, cost, and sustainability.
  1) Data are accessible only to the study team through an existing data license agreement between Temple University and the School District of Philadelphia. We do not anticipate the ability to preserve and share these data. 2) Transcripts will be de-identified and any potentially revealing information will be removed prior to sharing. 3) Survey data will be de-identified and any potentially revealing information will be removed prior to sharing.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available prior to publication of the first manuscript and will be made available open access until 10 years following the end of the trial period.

REFERENCES:
- [Derived] McLoughlin GM, Smith A, Dopp AR, Jones R, Martinez O, Kumanyika S, Yucel R, Brownson RC, Fisher JO. Using implementation mapping to optimize the impact of Universal School meals: a type III hybrid implementation-effectiveness study protocol. Implement Sci Commun. 2025 Oct 1;6(1):97. doi: 10.1186/s43058-025-00769-y. PMID 41034951